CLINICAL TRIAL: NCT03108677
Title: A Pilot Study of Circulating Exosome RNA as Diagnostic and Prognostic Markers in Lung Metastases of Primary High-Grade Osteosarcoma
Brief Title: Circulating Exosome RNA in Lung Metastases of Primary High-Grade Osteosarcoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Yuhui Shen, Ph.D., M.D., Ruijin Hospital
Other Study IDs: RJ2017NO13
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Lung Metastases; Osteosarcoma
Keywords: RNA profiling; Exosome; Lung Metastases; Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Samples with purified exosome RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- metastatic: For osteosarcoma patients with metastasis, collecting blood samples.
  Interventions: Other: Blood samples
- non-metastatic: For osteosarcoma patients without metastasis, collecting blood samples.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — 15 ml peripheral blood

SUMMARY:
The purpose of this study is to learn whether the profile of RNA from circulating exosomes can be used as a biomarker for lung metastases of primary high-grade osteosarcoma. Circulating exosomes plays roles in metastases in many kinds of cancer including osteosarcoma. By RNA profiling researchers may find lung metastases earlier than conventional work-up and predict the oncological outcomes.

DETAILED DESCRIPTION:
Investigators have performed a 4 patients pilot study under the oversight of hospital's ethics committee, and investigator found that the levels and mutations of circulating exosome RNA from patients with or without lung metastasis have significant differences. Then investigators wish to register this study to do a further research, in order to reveal the roles of circulating exosome RNA in metastases of osteosarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis by biopsy: primary high-grade osteosarcoma, including conventional osteosarcoma, telangiectatic osteosarcoma, small cell osteosarcoma, high-grade surface osteosarcoma.
* Tumor located in the extremities or pelvis.
* Age 12-60 years.
* No prior history of cancer and no prior treatment elsewhere.
* No prior history of chronic diseases including autoimmune disease, chronic infection, etc. which may interfere the level of circulating exosomes.

Exclusion Criteria:

* Initial misdiagnosis confirmed by specimen of definitive surgery.
* Applying target drugs in the period of treatment which may reduce tumor derived exosomes
* withdraw from the study for any reason

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with primary high-grade osteosarcoma aged 12-60.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Differences in the levels and mutations of circulating exosome RNA from patients with or without lung metastasis. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.

SECONDARY OUTCOMES:
Differences in the classic cell signal pathway mutations of circulating exosome RNA from patients with or without lung metastasis. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.
Differences in the therapeutic targets mutations of circulating exosome RNA from patients with or without lung metastasis. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.
The correlation between circulating exosome RNA mutation levels and 3-year disease-free survival (DFS), progression-free survival (PFS), lung metastases. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.
The correlation between specific circulating exosome RNA mutations and 3-year disease-free survival (DFS), progression-free survival (PFS), lung metastases. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.
The roles of circulating exosome micro-RNA mutations on regulation of circulating exosome RNA. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.
The mutations of circulating exosome RNA from patients without metastasis. | Before the neo-adjuvant chemotherapy, before the definitive surgery procedure, every 6 months after surgery. up to 3 years.
  Next generation sequencing will be performed to the whole RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Yuhui Shen, Ph.D., M.D., Principal Investigator — Ruijin Hospital; Weibin Zhang, Ph.D., M.D., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bao Q, Gong L, Wang J, Wen J, Shen Y, Zhang W. Extracellular Vesicle RNA Sequencing Reveals Dramatic Transcriptomic Alterations Between Metastatic and Primary Osteosarcoma in a Liquid Biopsy Approach. Ann Surg Oncol. 2018 Sep;25(9):2642-2651. doi: 10.1245/s10434-018-6642-z. Epub 2018 Jul 6. PMID 29981024